CLINICAL TRIAL: NCT00291161
Title: Partners in Dementia Care
Brief Title: Partners in Dementia Care: A Telephone Care Consultation Intervention Provided to Veterans in Partnership With Local Alzheimer's Association Chapters
Acronym: PDC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Benjamin Rose Institute (Other); Alzheimer's Association (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IIR 04-238
Record Dates: First submitted 2006-02-10; First posted 2006-02-13 (Estimated); Results first posted 2016-05-19 (Estimated); Last update posted 2016-05-19 (Estimated); Status verified 2016-05

CONDITIONS: Dementia; Alzheimer Disease
Keywords: Delivery of Health Care, Integrated; United States Department of Veterans Affairs; Dementia; Patient Care Management
MeSH Terms: conditions — Dementia; Alzheimer Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Partners in Dementia Care (Experimental): PDC is telephone-based care consultation intervention jointly delivered by care consultants in the VA and local Alzheimer's Association. The steps in care consultation included 1) Assessment of medical and non-medical care needs; 2) Development of a care plan that addresses needs of patients and caregivers; 3) on-going monitoring of the status, progress, and barriers encountered; and 4) Reassessment of care needs for patients and caregivers.
  PDC assisted families by: 1) providing disease-related education and information, 2) offering emotional support and coaching, 3) linking families to medical and non-medical services and resources, and 4) mobilizing and organizing the informal care network.
  Interventions: Behavioral: Partners in Dementia Care
- Usual Care (No Intervention): Patients and caregivers at the three control VA settings were given a packet of educational materials on dementia and usual-care community resources.

INTERVENTIONS:
Behavioral: Partners in Dementia Care — Partners in Dementia Care is facilitated by the VA Dementia care coordinator (VA DCC) that is with the study. The role of the VA DCC includes conducting initial assessments with the subject and caregiver that leads to:
  Arranging for further assessment or attention from VA health care system/providers about dementia related concerns or about co-morbid health issues; for example: VA driving evaluation, congestive heart failure medication adherence; Ensuring education is provided about particular health, safety issues; Following up with patient/caregiver on health promoting activities he/she is committed to do; and Sharing care plan actions/outcomes with other VA providers as agreed upon by patient.
  Arms: Partners in Dementia Care

SUMMARY:
Background: Partners in Dementia Care (PDC) is a care coordination and support service intervention for veterans with dementia and their family caregivers, delivered through partnerships between VA medical centers and local Alzheimer's Association Chapters. PDC was designed to be a feasible and practical intervention to integrate health, community, and support services. PDC has a standardized protocol for care coordination and support services, including guidelines for care plan assessment, care plan development and implementation, ongoing monitoring, and reassessment. It also offers a structured training curriculum for providers and an operations manual for uniform implementation.

Objectives: The primary objective was to test the impact of PDC on outcomes for veterans with dementia and family caregivers. Two specific research objectives and corresponding hypotheses were addressed: 1. To test the impact of PDC on three categories of outcomes: psychosocial well-being outcomes (patient and caregiver effects); health care service use (patient effects only); and health care cost (patient effects only). HI:PDC, compared to usual care, will improve psychosocial well-being for patients with dementia and their caregivers. H2:PDC, compared to usual care, will reduce health care service use for patients with dementia. H3:PDC is preferred to usual care based on cost-benefit analyses. H4:The PDC intervention will be more effective in improving psychosocial well-being and reducing health care service use for patients and caregivers dealing with more severe patient impairment (e.g., cognitive status, functional status, and level of problem behaviors). 2. To evaluate the impact of PDC on role and intra-psychic strains caused by dementia and its care (patient and caregiver effects). H5a:PDC, compared to usual care, will decrease patient role and intra-psychic strain. H5b:PDC, compared to usual care, will decrease caregiver role and intra-psychic strain. H6:The PDC intervention will be more effective in decreasing role and intra-psychic strains for patients and caregivers dealing with more severe patient impairment (e.g., cognitive status, functional status, and level of problem behaviors).

DETAILED DESCRIPTION:
Background:

Dementia affects the entire family by negatively impacting multiple domains including physical health, emotional health, social relationships, and legal and financial issues (Gurland, 1980; Kunik, Snow, Molinari, Menke, Souchek, Sullivan et al, 2003; Schulz, Visintainer, & Williamson, 1990; Wright, Clipp, & George, 1993). Particularly challenging is accessing the range of services needed to address the care needs of both the individual with dementia and the primary family caregiver. Common issues include: obtaining adequate diagnostic testing; understanding treatment options and medications; difficulties with memory and behavioral symptoms; and care- and illness-related strain (Mitnick, Leffler, & Hood, 2010). Additionally, many unmet care needs are the result of service fragmentation and inadequate communication among different medical providers, medical providers and consumers, and medical providers and community services (Reuben, Levin, Frank, 2009).

Built upon two prior studies: the Cleveland Alzheimer's Managed Care Demonstration (Bass, Clark, Looman, McCarthy, & Eckert, 2003) and the Chronic Care Networks for Alzheimer's Disease (CCN/AD) (Maslow & Bass, 2003; Maslow & Selstad, 2001), PDC was a 5-year research investigation that tested the effectiveness of a telephone-based, innovative care-coordination intervention designed to address the unmet care needs of Veterans with dementia and their family caregivers across all dementia stages. PDC was implemented through formal partnerships between the VA medical centers and local Alzheimer's Association (AA) chapters. Essential features of PDC included: 1) formal partnerships between VA medical centers and Alzheimer's Association Chapters; 2) a multidimensional assessment and treatment approach, 3) ongoing monitoring and long-term relationships with families; and 4) a computerized information system to guide service delivery and fidelity monitoring. For a complete description of the PDC intervention protocol please see Judge, Bass, Snow, Wilson, Morgan, Looman, McCarthy, and Kunik (2010).

Objectives:

The primary objective of this investigation is to rigorously test the impact of PDC on a number of outcomes for Veterans with dementia, family caregivers, and healthcare providers. Within VA Medical Centers, the focus will be on improving dementia care in primary care clinics, including geriatrics.

Two specific research objectives and corresponding hypotheses will be addressed:

1. To test the impact of PDC on three categories of outcomes: psychosocial well-being outcomes (patient and caregiver effects); healthcare service use (patient effects only); and health care cost (patient effects only).

   Hypothesis 1: PDC, compared with usual care, will improve psychosocial well-being, including depression, health status, adequacy of care, and quality of care for patients with dementia and their caregivers.

   Hypothesis 2: PDC, compared with usual care, will reduce healthcare service use for patients with dementia, including hospital admissions, emergency department visits, nursing home admissions, and physician visits.

   Hypothesis 3: PDC is preferred to usual care, based on cost-effectiveness and cost-benefit analyses.

   Hypothesis 4: The PDC intervention will be more effective than usual care in improving psychosocial well-being and reducing health care service use for patients and caregivers dealing with more severe patient impairment (e.g., cognitive status, functional status, and level of problem behaviors).
2. To evaluate the impact of PDC on role and intra-psychic strains caused by dementia and its care (patient and caregiver effects).

Hypothesis 5a: PDC, compared with usual care, will decrease patient role and intra-psychic strain, including embarrassment about the illness, emotional strain, relationship strain, and social isolation.

Hypothesis 5b: PDC, compared with usual care, will decrease caregiver role and intra-psychic strain, including role captivity, work care-related strain, relationship strain, emotional and physical health deterioration, and caregiving efficacy.

Hypothesis 6: The PDC intervention will be more effective than usual care in decreasing role and intra-psychic strains for patients and caregivers dealing with more severe patient impairment (e.g., cognitive status, functional status, and level of problem behaviors).

Methods:

The proposed study was a 55-month, controlled trial of PDC. The project was conducted at two intervention sites and three comparison sites matched on organizational, provider, and patient characteristics.

Partners in Dementia Care was compared to usual care. Both groups received educational materials about dementia at the start.

PDC Intervention The Chronic Care Model (Bodenheimer, Wagner, & Grumbach, 2002; Bodenheimer, Wagner, & Grumbach, 2002) was used as an overarching framework to implement PDC and included the following components: 1) Formal linkages between medical centers (the VA) and community agencies (the Alzheimer's Association); 2) Organizational support from key leaders and broad-based training about PDC; 3) Delivery system redesign and decision support systems; 4) Self-management of dementia as outlined by the PDC intervention protocol; 5) The development of the PDC Care Coordination Information System (CCIS) as the clinical information system.

PDC had four primary ways of assisting families: 1) providing disease-related education and information; 2) offering emotional support and coaching; 3) linking families to medical and non-medical services and resources; and 4) mobilizing and organizing the informal care network. Two key staff members implemented the intervention: a VA Dementia Care Coordinator (VA DCC) in VA medical centers and an Alzheimer's Association Care Consultant (AA CC) in Alzheimer's Association Chapters. VA DCCs primarily focused on veterans' medical and non-medical needs and assisted families with effectively using VA resources; AA CCs primarily focused on needs of informal caregivers such as care-related strain and accessing non-VA resources. The intervention protocol consisted of: 1) Assessment of Care Needs across medical and non-medical care issues that addressed 23 domains for Veterans and 14 domains for caregivers; 2) Development of Care Goals that matched the priorities of Veterans and caregivers; 3) Development of Action Steps which were concrete behavioral tasks intended to help families move toward goal achievement (e.g., individual responsible for completing each task, expected completion date); 4) On-going Monitoring of Action Steps on a regular basis to ensure timely completion of tasks, address potential barriers, modify or add action steps, and identify new goals.

Analytic Plan With one exception, measures of "objective" characteristics, including community and support-service use, service knowledge, number of informal helpers, and Veterans' impairments, were based on information reported by caregivers. The one exception was a measure of impairment based on scores from a standardized mental status test that was administered to Veterans over the telephone (i.e., the Blessed Orientation-Memory-Concentration Test; Katzman et al., 1983). Additionally, a small number of Veterans (approximately 5%) with mild dementia did not have a caregiver; "objective" characteristics for these individuals were self-reported by the Veteran. Information used to construct measures of "subjective" characteristics, such as feelings about or perceptions of the quality of care and care-related strain, came directly from the individual whose feelings or perceptions were being represented.

ELIGIBILITY:
Inclusion Criteria:

* Dementia Diagnosis
* veteran
* reside outside of a long-term care facility
* live within local Alzheimer Association chapter service of Houston, Oklahoma City, Boston, or Providence

Exclusion Criteria:

* Live in long-term care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 994 (Actual)
Dates: Start 2006-12; Primary Completion 2010-09 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark E Kunik, MD MPH, Principal Investigator — Michael E. DeBakey VA Medical Center
Locations (6):
- United States (6):
  - VA Boston Health Care System, Jamaica Plain, Boston, Massachusetts
  - VA Boston Healthcare System, Brockton Campus, Brockton, Massachusetts
  - Oklahoma City, OK, Oklahoma City, Oklahoma
  - VA Medical Center, Providence, Providence, Rhode Island
  - Beaumont VA Outpatient Clinic, Beaumont, Texas
  - Michael E DeBakey VA Medical Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Shrestha S, Judge KS, Wilson NL, Moye JA, Snow AL, Kunik ME. Utilization of legal and financial services of partners in dementia care study. Am J Alzheimers Dis Other Demen. 2011 Mar;26(2):115-20. doi: 10.1177/1533317510394156. Epub 2011 Jan 13. PMID 21233136
- [Background] Judge KS, Bass DM, Snow AL, Wilson NL, Morgan R, Looman WJ, McCarthy C, Kunik ME. Partners in dementia care: a care coordination intervention for individuals with dementia and their family caregivers. Gerontologist. 2011 Apr;51(2):261-72. doi: 10.1093/geront/gnq097. Epub 2011 Jan 17. PMID 21242317
- [Background] Bradford A, Upchurch C, Bass D, Judge K, Snow AL, Wilson N, Kunik ME. Knowledge of documented dementia diagnosis and treatment in veterans and their caregivers. Am J Alzheimers Dis Other Demen. 2011 Mar;26(2):127-33. doi: 10.1177/1533317510394648. Epub 2011 Jan 27. PMID 21273206
- [Background] Weber SR, Pirraglia PA, Kunik ME. Use of services by community-dwelling patients with dementia: a systematic review. Am J Alzheimers Dis Other Demen. 2011 May;26(3):195-204. doi: 10.1177/1533317510392564. Epub 2011 Jan 27. PMID 21273207
- [Background] Shub D, Bass DM, Morgan RO, Judge KS, Snow AL, Wilson NL, Walder A, Murry B, Kunik ME. Irritability and social isolation in dementia patients with and without depression. J Geriatr Psychiatry Neurol. 2011 Dec;24(4):229-34. doi: 10.1177/0891988711427039. PMID 22228830
- [Background] Bass DM, Judge KS, Snow AL, Wilson NL, Looman WJ, McCarthy C, Morgan R, Ablorh-Odjidja C, Kunik ME. Negative caregiving effects among caregivers of veterans with dementia. Am J Geriatr Psychiatry. 2012 Mar;20(3):239-47. doi: 10.1097/JGP.0b013e31824108ca. PMID 22251867
- [Background] Bejjani C, Snow AL, Judge KS, Bass DM, Morgan RO, Wilson N, Walder A, Looman WJ, McCarthy C, Kunik ME. Characteristics of Depressed Caregivers of Veterans With Dementia. Am J Alzheimers Dis Other Demen. 2015 Nov;30(7):672-8. doi: 10.1177/1533317512461555. Epub 2012 Oct 14. PMID 23070578
- [Background] Godwin KM, Morgan RO, Walder A, Bass DM, Judge KS, Wilson N, Snow AL, Kunik ME. Predictors of Inpatient Utilization among Veterans with Dementia. Curr Gerontol Geriatr Res. 2014;2014:861613. doi: 10.1155/2014/861613. Epub 2014 May 29. PMID 24982674
- [Background] Ng S, Morgan RO, Walder A, Biswas J, Bass DM, Judge KS, Snow AL, Wilson N, Kunik ME. Functional Decline Predicts Emergency Department Use in Veterans With Dementia. Am J Alzheimers Dis Other Demen. 2014 Jun;29(4):362-71. doi: 10.1177/1533317513518655. Epub 2014 Jan 9. PMID 24413540
- [Result] Steiger-Gallagher K, Bass DM, Judge KS, Snow L, Wilson NL, Morgan RO, Walder A, Kunik ME. Satisfaction with dementia care. Federal practitioner : for the health care professionals of the VA, DoD, and PHS. 2012 Apr 1; 29(4):33-40.
- [Result] Bass DM, Judge KS, Snow AL, Wilson NL, Morgan R, Looman WJ, McCarthy CA, Maslow K, Moye JA, Randazzo R, Garcia-Maldonado M, Elbein R, Odenheimer G, Kunik ME. Caregiver outcomes of partners in dementia care: effect of a care coordination program for veterans with dementia and their family members and friends. J Am Geriatr Soc. 2013 Aug;61(8):1377-86. doi: 10.1111/jgs.12362. Epub 2013 Jul 19. PMID 23869899
- [Result] Bass DM, Judge KS, Snow AL, Wilson NL, Morgan RO, Maslow K, Randazzo R, Moye JA, Odenheimer GL, Archambault E, Elbein R, Pirraglia P, Teasdale TA, McCarthy CA, Looman WJ, Kunik ME. A controlled trial of Partners in Dementia Care: veteran outcomes after six and twelve months. Alzheimers Res Ther. 2014 Feb 28;6(1):9. doi: 10.1186/alzrt242. eCollection 2014. PMID 24764496
- [Result] Morgan RO, Bass DM, Judge KS, Liu CF, Wilson N, Snow AL, Pirraglia P, Garcia-Maldonado M, Raia P, Fouladi NN, Kunik ME. A break-even analysis for dementia care collaboration: Partners in Dementia Care. J Gen Intern Med. 2015 Jun;30(6):804-9. doi: 10.1007/s11606-015-3205-x. Epub 2015 Feb 10. PMID 25666216
- [Derived] Bass DM, Judge KS, Maslow K, Wilson NL, Morgan RO, McCarthy CA, Looman WJ, Snow AL, Kunik ME. Impact of the care coordination program "Partners in Dementia Care" on veterans' hospital admissions and emergency department visits. Alzheimers Dement (N Y). 2015 Apr 17;1(1):13-22. doi: 10.1016/j.trci.2015.03.003. eCollection 2015 Jun. PMID 29854922
- See also: AHRQ Healthcare Innovations Exchange — https://innovations.ahrq.gov/profiles/partnership-supports-patients-dementia-and-their-caregivers-through-care-coordinator-team

RESULTS

PARTICIPANT FLOW:
Groups:
- Veterans: Partners in Dementia Care Intervention: A two-person care coordinator team, one based at the VA and one based at the Alzheimer Association, provided telephone-based support to patients with dementia and their caregivers over a 12-month period. The team addressed medical and nonmedical needs through education, coaching, linkages to needed resources, and mobilization of an informal care network. The program consisted of an upfront assessment, development of care goals and action steps, and ongoing monitoring and intervention by the two coordinators, who communicated with each other regularly.
- Veterans: Usual Care Comparison: Patients and caregivers were provided usual care and an educational booklet on dementia
- Caregivers: Partners in Dementia Care Intervention: Caregivers for Veterans assigned to the Partners in Dementia Care Intervention
- Caregivers: Usual Care Comparison: Caregivers of the Veterans assigned to the Usual Care Comparison
Period: Overall Study
Arm/Group | Veterans: Partners in Dementia Care Intervention | Veterans: Usual Care Comparison | Caregivers: Partners in Dementia Care Intervention | Caregivers: Usual Care Comparison
Started | 316 | 192 | 299 | 187
Completed | 235 | 134 | 206 | 122
Not Completed | 81 | 58 | 93 | 65

BASELINE CHARACTERISTICS:
Groups:
- Veterans-PDC Group: Veterans with diagnosed dementia receiving the PDC Intervention
- Veterans-Usual Care Comparison Group: Veterans with diagnosed dementia receiving educational materials and usual care
- Caregivers-PDC Group: Caregivers to veterans with diagnosed dementia receiving the PDC Intervention
- Caregivers-Usual Care Comparison Group: Caregivers to veterans with diagnosed dementia receiving educational materials and usual care
- Total: Total of all reporting groups
Arm/Group | Veterans-PDC Group | Veterans-Usual Care Comparison Group | Caregivers-PDC Group | Caregivers-Usual Care Comparison Group | Total
Number analyzed (Participants) | 316 | 192 | 299 | 187 | 994
Age, Continuous [Mean (Standard Deviation); unit: years]
  Age of Veterans | 79.4 (8.2) | 80.7 (6.2) | NA (NA) — Age of veterans measured separate from age of caregivers | NA (NA) — Age of veterans measured separate from age of caregivers | 79.9 (7.6)
  Age of Caregivers | NA (NA) — Age of veterans measured separate from age of caregivers | NA (NA) — Age of veterans measured separate from age of caregivers | 68.0 (12.6) | 70.8 (11.4) | 69.1 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 3 | 283 | 178 | 475
  Male | 305 | 189 | 16 | 9 | 519
Race/Ethnicity, Customized [Number; unit: participants]
  White nonhispanic | 234 | 178 | 222 | 170 | 804
  Black nonhispanic | 64 | 11 | 56 | 14 | 145
  Hispanic | 12 | 0 | 16 | 0 | 28
  Other | 6 | 3 | 5 | 3 | 17
Number of Caregivers Who were Spouses [Number; unit: participants] — Was only collected for Caregiver groups
  participants
    Caregivers who were spouses | NA — Was only collected for Caregiver groups | NA — Was only collected for Caregiver groups | 204 | 149 | NA — Total not calculated because data are not available (NA) in one or more arms.
    Caregivers who were not spouses | NA — Was only collected for Caregiver groups | NA — Was only collected for Caregiver groups | 95 | 38 | NA — Total not calculated because data are not available (NA) in one or more arms.

OUTCOME MEASURES:

1. Primary Outcome: Caregiver Outcomes
Description: The following outcomes were measured in Caregivers via scales administered to each caregiver: Unmet need (range=0 to 39, higher meaning more unmet needs); Role captivity (range=0-9, higher indicating greater role captivity); Physical health strain (range=0-9, higher indicating greater health strain); Relationship strain (range=0-18, higher indicating greater relationship strain); Depression (range=0-22, higher indicating greater depression); Caregiver support service use (the number of support services utilized, 0-2); Number of informal helpers (range=0-50, higher indicating more informal helpers)
Time Frame: Baseline and at six months
Population: Data were collected for caregivers only
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Caregivers: Partners in Dementia Care Intervention: A two-person care coordinator team, one based at the VA and one based at the Alzheimer Association, provided telephone-based support to patients with dementia and their caregivers over a 12-month period. The team addressed medical and nonmedical needs through education, coaching, linkages to needed resources, and mobilization of an informal care network. The program consisted of an upfront assessment, development of care goals and action steps, and ongoing monitoring and intervention by the two coordinators, who communicated with each other regularly.
- Caregivers: Usual Care Comparison: Patients and caregivers were provided usual care and an educational booklet on dementia
Arm/Group | Caregivers: Partners in Dementia Care Intervention | Caregivers: Usual Care Comparison
Number analyzed (Participants) | 299 | 187
units on a scale
  Unmet need at Baseline | 18.6 (11.8) | 14.5 (11.2)
  Unmet need at Six months | 10.0 (9.9) | 10.5 (10.0)
  Role Captivity at baseline | 3.7 (1.6) | 3.5 (1.4)
  Role Captivity at 6 months | 3.6 (1.6) | 3.2 (1.6)
  Physical Health Strain at Baseline | 3.7 (1.6) | 3.6 (1.3)
  Physical Health Strain at 6 months | 3.5 (1.4) | 3.6 (1.5)
  Relationship Strain at Baseline | 7.2 (2.5) | 6.8 (2.1)
  Relationship Strain at 6 months | 7.0 (2.6) | 6.3 (2.3)
  Caregiver Support Service use at baseline | .4 (.7) | .4 (.7)
  Caregiver support service at 6 months | .7 (.7) | .5 (.7)
  Depression at baseline | 4.5 (3.9) | 4.0 (2.9)
  Depression at 6 months | 4.7 (3.9) | 5.0 (4.1)
  Number of informal helpers at baseline | 4.3 (4.8) | 4.3 (5.1)
  Number of informal helpers at 6 month | 4.7 (5.8) | 4.8 (9.1)

2. Primary Outcome: Veteran Outcomes
Description: The following outcomes were measured for veterans via scales administered to each veteran: Unmet need (range=0 to 24, higher meaning more unmet needs); Embarrassment about memory problems (range=0-3, higher indicating greater embarrassment); Isolation (range=0-4, higher indicating greater isolation); Relationship strain (range=0-4, higher indicating greater relationship strain); Depression (range=0-11, higher indicating greater depression).
Time Frame: Baseline - six months
Population: Data were collected for veterans who could be interviewed only.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Partners in Dementia Care Intervention: A two-person care coordinator team, one based at the VA and one based at the Alzheimer Association, provided telephone-based support to patients with dementia and their caregivers over a 12-month period. The team addressed medical and nonmedical needs through education, coaching, linkages to needed resources, and mobilization of an informal care network. The program consisted of an upfront assessment, development of care goals and action steps, and ongoing monitoring and intervention by the two coordinators, who communicated with each other regularly.
- Usual Care Comparison: Patients and caregivers were provided usual care and an educational booklet on dementia
Arm/Group | Partners in Dementia Care Intervention | Usual Care Comparison
Number analyzed (Participants) | 152 | 103
units on a scale
  Embarrassment about memory problems at baseline | 1.02 (1.19) | .89 (1.08)
  Embarrassment about memory problems at 6 months | .82 (1.09) | .91 (1.10)
  Depression at baseline | 2.68 (2.44) | 2.19 (2.10)
  Depression at 6 months | 2.52 (2.59) | 2.37 (2.34)
  Unmet need at baseline | 7.00 (6.93) | 5.44 (6.00)
  Unmet need at 6 months | 5.05 (6.14) | 4.40 (5.58)
  Isolation at baseline | 1.38 (1.49) | 1.06 (1.30)
  Isolation at 6 months | 1.13 (1.39) | 1.09 (1.37)
  Relationship strain at baseline | .46 (1.04) | .38 (.87)
  Relationship strain at 6 months | .49 (1.02) | .32 (.79)

ADVERSE EVENTS:
Description: Adverse Events only assessed for Veterans
Arm/Group | Veterans-PDC Group | Veterans-Usual Care Comparison Group
Serious Adverse Events (participants affected / at risk) | 0/316 | 0/192
Other Adverse Events (participants affected / at risk) | 0/316 | 0/192

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No